CLINICAL TRIAL: NCT02276391
Title: Bioequivalence of Telmisartan Administrated in Two Different Ways: Either in Telmisartan 80 mg/HCTZ 12.5 mg Fixed-dose Combination Tablet or as Two Telmisartan 40 mg Tablets (an Open-label, Randomised, Single-dose, Four-period Replicated Crossover Study)
Brief Title: Bioequivalence of Telmisartan as Telmisartan 80 mg/HCTZ 12.5 mg Fixed-dose Combination Tablet or as Two Telmisartan 40 mg Tablets in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 502.571
Record Dates: First submitted 2014-10-27; First posted 2014-10-28 (Estimated); Last update posted 2014-10-28 (Estimated); Status verified 2014-10

CONDITIONS: Healthy
MeSH Terms: interventions — Telmisartan

ARMS (2):
- Telmisartan/HCTZ fixed-dose combination (Experimental)
  Interventions: Drug: Telmisartan/HCTZ combination
- Telmisartan (Active Comparator)
  Interventions: Drug: Telmisartan

INTERVENTIONS:
Drug: Telmisartan/HCTZ combination
  Arms: Telmisartan/HCTZ fixed-dose combination
Drug: Telmisartan
  Arms: Telmisartan

SUMMARY:
To establish bioequivalence of telmisartan orally administrated in two different ways: either with a telmisartan 80 mg/hydrochlorothiazide (HCTZ) 12.5 mg fixed-dose combination tablet or with two telmisartan 40 mg tablets

ELIGIBILITY:
Inclusion Criteria:

Healthy Japanese males according to the following criteria:

1. Based upon a complete medical history, including the physical examination, vital signs (blood pressure (BP), pulse rate (PR), body temperature), 12-lead ECG (electrocardiogram), clinical laboratory tests
2. Age ≥20 and Age ≤35 years
3. Body weight ≥50 kg
4. Body Mass Index (BMI) ≥18.0 and BMI ≤25.0 kg/m2
5. Signed and dated written informed consent prior to admission to the study in accordance with Good Clinical Practice (GCP) and the local legislation.

Exclusion Criteria:

1. Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
2. Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
3. Chronic or relevant acute infections
4. Any clinical relevant findings of the laboratory test deviating from normal
5. Positive result for either hepatitis B surface (HBs) antigen, anti hepatitis C virus (HCV) antibodies, syphilitic test or human immunodeficiency virus (HIV) test
6. History of surgery of gastrointestinal tract (except appendectomy)
7. History of relevant orthostatic hypotension, fainting spells or blackouts
8. Known hypersensitivity to any component of the formulation (telmisartan and hydrochlorothiazide), or to any other angiotensin II receptor blocker (ARBs), any other thiazides, or thiazide derivatives (e.c. sulfonamide derivatives like a chlorthalidone)
9. History of hepatic dysfunction (e.g. biliary cirrhosis, cholestasis)
10. History of serious renal dysfunction
11. History of bilateral renal artery stenosis or renal artery stenosis in a solitary kidney
12. History of cerebrovascular disorder
13. History of hyperkalemia
14. History of impaired glucose tolerance
15. History of hypokalemia
16. History of hyperuricemia
17. Salt restriction therapy
18. Intake of drugs with a long half-life (≥24 hours) within at least one month or less than 10 half-lives of the respective drug prior to administration or during the trial
19. Use of drugs which might reasonably influence the results of the trial based on the knowledge at the time of protocol preparation within 7 days prior to administration or during the trial
20. Participation in another trial with an investigational drug within 4 months or 6 half-lives of the investigational drug prior to administration
21. Smoker (≥20 cigarettes /day))
22. Alcohol abuse (60 g or more ethanol/day: ex. 3 middle-sized bottles of beer, 3 gous (equivalent to 540 mL) of sake)
23. Drug abuse
24. Blood donation (more than 100 mL within 4 weeks prior to administration or during the trial)
25. Excessive physical activities (within 1 week prior to administration or during the trial)
26. Intake of alcohol within 2 days prior to administration
27. Inability to comply with dietary regimen of study centre
28. Inability to refrain from smoking on trial days
29. Subjects judged to be inappropriate by the investigator or the sub-investigator

Ages: 20 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2008-07; Primary Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
AUC0-tz (area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the time of the last quantifiable data point) | Up to 72 hours after drug administration
Cmax (maximum measured concentration of the analyte in plasma) | Up to 72 hours after drug administration

SECONDARY OUTCOMES:
AUC0-∞ (area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity) | Up to 72 hours after drug administration
tmax (time from dosing to the maximum measured concentration of the analyte in plasma) | Up to 72 hours after drug administration
λz (terminal rate constant of the analyte in plasma) | Up to 72 hours after drug administration
t1/2 (terminal half-life of the analyte in plasma) | Up to 72 hours after drug administration
MRTpo (mean residence time of the analyte in the body after po administration) | Up to 72 hours after drug administration
Number of participants with clinically significant findings in physical examination | Up to 72 hours after last drug administration
Number of participants with clinically significant findings in vital signs | Up to 72 hours after last drug administration
Number of participants with clinically significant findings in 12-lead ECG (electrocardiogram) | Up to 72 hours after last drug administration
Number of participants with clinically significant findings in clinical laboratory parameters | Up to 72 hours after last drug administration
Number of participants with adverse events | Up to 72 hours after last drug administration